CLINICAL TRIAL: NCT04096521
Title: Serum Folic Acid Status, Genotyping MTHFR 677C-->T of the Mother and Serum Folic Acid Status, DNA Methylation of IGF2 Gene of the Children: East Jakarta Cohort Study
Brief Title: Serum Folic Acid Status, Genotyping MTHFR 677C-->T, Plasma Homocysteine, DNA Methylation of IGF2 Gene and Microbiota of the Children: Mother-Children Cohort Study
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Collaborators: Ministry of Research and Higher Education of Republic Indonesia (Unknown); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lestari Octavia, MSc, Indonesia University
Other Study IDs: 0420/UN2.F1/ETIK/2018
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Folic Acid Deficiency
Keywords: serum folic acid; genotyping; dna methylation of IGF2; East Jakarta Cohort Study; mother-children
MeSH Terms: conditions — Folic Acid Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA isolated from the whole blood using standardized equipment and procedure of blood taking.
  DNA obtained from mother-children of the participant in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- East Jakarta Cohort Study: One group included in the study was originated from mothers who participated in the first data collection pregnancy. The follow-up study included mothers and their children born as the subject in the follow-up in the study. This study also includes peer of the subjects that lived in the same neighbourhood since the first cohort study and have children in the same age with cohort participant

SUMMARY:
This study is part of the East Jakarta Cohort Study to assess the current micronutrient status of the mothers and their children. The study also includes the assessment of genotyping of MTHFR 677C-->T of the mother and DNA methylation of IGF2 gene of the children.

DETAILED DESCRIPTION:
The initial study recruited 315 mothers in the public health centre and one district hospital in East Jakarta. The follow-up study is able to re-visit the 127 of them. This also includes 127 peers of the subject that lives in the same neighbourhood. The design of the study is case-cohort design, part study of the existing cohort. The assessment of the follow-up study includes the mother and the children born in the initial study. Anthropometric measurement, socioeconomic data from a structured questionnaire, biomarker assessment, blood pressure were obtained from the subjects.

ELIGIBILITY:
Inclusion Criteria:

* participant in the previous study
* apparently healthy
* data complete
* voluntarily to participate

Exclusion Criteria:

* not complete data
* migrate
* refuse to participate in the study

Ages: 3 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: In 2014, the pregnant mothers in 10 public health centre and one sub-district hospital in East Jakarta were recruited in the study. They were in the third trimester gestation period, receive iron-folic acid supplementation and ANC. In 2018, the repeated collection was conducted to collect follow-up data. We also include peer of the subjects that lived in the same neighbourhood since the first cohort study and have children in the same age with cohort participant
Sampling Method: Non-Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2019-03-16 (Actual)

PRIMARY OUTCOMES:
Serum folic acid status | December 2018 - March 2019
  The measurement of serum folic acid status is using LC-MS/MS
Genotyping MTHFR 677C-->T | December 2018 - March 2019
  The assessment of MTHFR 677C-->T using Real Time PCR
DNA methylation of IGF2 gene | December 2018 - March 2019
  DNA methylation of IGF2 gene using pyrosequencing method

SECONDARY OUTCOMES:
Serum Homocysteine | December 2018-March 2019
  The measurement of serum homocysteine using Electrochemiluminescen
Serum Adiponectin | December 2018-March 2019
  The measurement of serum adiponection using electrochemiluminescence
Blood pressure | December 2018-March 2019
  The blood pressure measurement using semi automatic device (Omron HBP1300)

OTHER OUTCOMES:
Nutritional status assessment | September 2018-December 2018
  Using antrhopometric measurement, using SECA for weight measurement, Shorrboard for height and standardized plastic tape for mid upper arm circumference.

CONTACTS AND LOCATIONS:
Overall Officials: Rina RA Agustina, Doctoral, Study Director — Indonesia University
Locations (1):
- Universitas Indonesia, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No
I will not share the IPD of the subject participated due to consent issue

REFERENCES:
- See also: The maternal folic acid supplementation results strengthen the link between folic acid supplementation during later pregnancy and epigenetic changes and identify a novel mechanism for regulation of ZFP57. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6380035